CLINICAL TRIAL: NCT04772404
Title: Repercussion of the COVID-19 Pandemic on Physical Activity, Psychological State and Sleep
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator; PT; PhD, Universidad de Granada
Other Study IDs: DF0094UG
Record Dates: First submitted 2021-02-12; First posted 2021-02-26 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-19 outbreak in our environment has caused significant changes in the population. The main objective of this research project is to evaluate the level of physical activity, psychological state and sleep during the COVID-19 pandemic in different populations.

ELIGIBILITY:
Inclusion Criteria:

• Healthy people

Exclusion Criteria:

* Cognitive impairment.
* Diagnose of autism spectrum disorder or severe intellectual disability
* Physical or functional impairment that limits the performance of evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy people
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-07 (Actual); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Knowledge of COVID | Baseline
  Questionnaire to evaluate the knowledge about COVID-19. It includes 12 items. Patients have to answer true/false. Higher puntuation indicates better knowledge results.
Fear of COVID-19 Scale | Baseline
  Bangla fear of COVID (FCV19-S): It is a questionnaire that assesses the fear of COVID-19. It consists of 7 items scored on a 5-item Likert scale. The higher the score, the more fear.
COVID-19 Anxiety Scale (CAS) | Baseline
  Coronavirus anxiety scale (CAS): It is a scale that measures the anxiety generated by COVID-19 in the last two weeks. It presents 5 items and a score> 9 indicates dysfunctional anxiety associated with the pandemic.
COVID Stress Scales | Baseline
  COVID stress scale (CSS): is a 36-item COVID Stress Scale (CSS) to measure these features, as they pertain to COVID-19. The CSS were developed to better understand and assess COVID-19-related distress. The scales were intentionally designed so they could be readily adapted for future pandemics.
Burn-Out de Maslach Inventory | Baseline
  The Maslach Burnout Inventory (MBI) is a psychological assessment instrument comprising 22 symptom items pertaining to occupational burnout
Steps per day | Baseline
  Accelerometer
International physical activity questionnaire | Baseline
  The International Physical Activity Questionnaire (IPAQ) was developed to measure health-related physical activity (PA) in populations. Higher scores indicates higher physical activity levels.
Barriers to being active quiz | Baseline
  Barriers to being active quiz (BBAQ-21): It is a questionnaire that consists of 21 items. This questionnaire was aimed at ascertaining perception of barriers against engaging in PA.
Questionnaire of the transtheoretical model of change of physical exercise | Baseline
  Questionnaire of the transtheoretical model of change of physical exercise (QTMCPE): It is made up of 22 items for people who are not physically active and 9 items for physically active people. It is a Likert-type scale that measures from 1 to 5.
Hospital Anxiety and Depression Scale | Baseline
  Anxiety and depression will be assessed with the Hospital Anxiety and Depression Scale (HADS) . This scale is composed of 14 items divided into two subscales, 7 items of anxiety and 7 items of depression, involving higher values worse psycho-emotional state.
Connor-Davidson Resilience Scale | Baseline
  Connor-Davidson Resilience Scale (CD-RISC) was used to measure resilience. It consists of 10 items which form five factors. Respondents are asked to answer on a five-point Likert scale (0 = totally disagree to 4 = totally agree).
COPE-28 | Baseline
  The Brief-COPE is a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. "Coping" is defined broadly as an effort used to minimize distress associated with negative life experiences.
Pittsburgh Sleep Quality Index | Baseline
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances in the previous month.
Morningness-eveningness questionnaire (MEQ) | Baseline
  Morningness-Eveningness Questionnaire: Consisting of 19 items, the scale was developed to assess individual differences in morningness and eveningness - the degree to which respondents are active and alert at certain times of day. Scale items query preferences in sleep and waking times, and subjective "peak" times at which respondents feel their best.
Epworth sleepiness Scale | Baseline
  The ESS asks the respondent to rate on a 4-point scale (0-3) their usual chances of having dozed off or fallen asleep while engaged in eight different activities that differ widely in their somnificity.
Insomnia severity index | Baseline
  Insomnia severity index: It consists of 24 questions that measure sleep disturbances along dimensions: subjective sleep quality, sleep latency (LS), duration, efficiency, sleep disorders, use of sleep medication, and daytime dysfunction. The evaluation is based on the answers obtained from the previous month.

SECONDARY OUTCOMES:
EuroQoL-5D | Baseline
  The perception of the level of health and the quality of life were evaluated with the questionnaire European Quality of
  Life-5 Dimensions (EQ-5D). It is composed of 2 parts in which health status is assessed:
  Descriptive system: It consists on 5 dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Patients classify their health status in 3 severity levels: having no problems, having some or moderate problems, being unable to do/having extreme problems.
  Visual Analog Scale, by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status)
Charlson Comorbidity Index | Baseline
  Charlson Comorbidity Index predicts the ten-year mortality for a patient who may have a range of comorbid conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, Granada, Spain

IPD SHARING:
Plan to Share IPD: No